CLINICAL TRIAL: NCT03595592
Title: Atezolizumab, Pertuzumab and Trastuzumab With Chemotherapy as Neoadjuvant Treatment of HER2 Positive Early High-risk and Locally Advanced Breast Cancer (APTneo)
Brief Title: Neoadjuvant Treatment of HER2 Positive Early High-risk and Locally Advanced Breast Cancer
Acronym: APTneo
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FM-17-B01; 2017-000981-31 (EudraCT Number)
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Invasive Breast Cancer
Keywords: Unilateral, HER2 positive
MeSH Terms: interventions — Trastuzumab; pertuzumab; Carboplatin; Paclitaxel; Doxorubicin; Cyclophosphamide; atezolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Parallel randomization to the study arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HPCT (Active Comparator): Patients will receive a combination of trastuzumab, pertuzumab, carboplatin and paclitaxel as neoadjuvant therapy for 6 cycles every 3 weeks. Trastuzumab (H) will be delivered on day 1 at the dose of 8 mg/kg loading dose i.v., then 6 mg/kg i.v. Pertuzumab (P) will be delivered on day 1 at the dose of 840 mg loading dose i.v., then 420 mg i.v. Carboplatin (C) will be administered at AUC 2 i.v. on day 1 and day 8. Paclitaxel (T) will be given at 90 mg/m2 i.v. on day 1 and day 8. Definite surgery will be performed not later than 4 weeks after the last dose of neoadjuvant therapy. Trastuzumab and pertuzumab will then be delivered for 12 additional cycles as adjuvant therapy.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Surgery
- ACy followed by HPCT and atezolizumab (Experimental): Patients will receive a combination of doxorubicin (A, 60 mg/m2 i.v.), cyclophosphamide (C, 600 mg/m2 i.v.) and atezolizumab (1200 mg i.v.) on day 1 every 3 week for 3 cycles. Subsequently they will be given trastuzumab on day 1 (H, at the loading dose of 8 mg/kg i.v. then 6 mg/kg i.v.), pertuzumab on day 1 (P, at the loading dose of 840 mg .v., then 420 mg i.v.), carboplatin (C) at AUC 2 i.v. on day 1 and day 8, paclitaxel (T) at 90 mg/m2 i.v. on day 1 and day 8, and atezolizumab 1200 mg i.v. on day 1 for 3 cycles every 3 weeks. Definite surgery will be performed not later than 4 weeks after the last dose of neoadjuvant therapy. Trastuzumab and pertuzumab will then be delivered for 15 additional cycles and atezolizumab for 12 additional cycles as adjuvant therapy.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Atezolizumab; Procedure: Surgery
- HPCT and atezolizumab (Experimental): Patients will receive a combination of trastuzumab, pertuzumab, carboplatin, paclitaxel and atezolizumab as neoadjuvant therapy for 6 cycles every 3 weeks. Trastuzumab (H) will be delivered on day 1 at the dose of 8 mg/kg loading dose i.v., then 6 mg/kg i.v. Pertuzumab (P) will be delivered on day 1 at the dose of 840 mg loading dose i.v., then 420 mg i.v. Carboplatin (C) will be administered at AUC 2 i.v. on day 1 and day 8; paclitaxel (T) will be given at 90 mg/m2 i.v. on day 1 and day 8; atezolizumab at the dose of 1200 mg i.v. on day 1. Definite surgery will be performed not later than 4 weeks after the last dose of neoadjuvant therapy. Trastuzumab, pertuzumab and atezolizumab will then be delivered for 12 additional cycles as adjuvant therapy.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Atezolizumab; Procedure: Surgery

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be given i.v. on day 1 every 3 weeks in arms HPCT, ACy followed by HPCT and atezolizumab and in arm HPCT and atezolizumab
  Other Names: Herceptin
Drug: Pertuzumab — Pertuzumab will be given i.v. on day 1 every 3 weeks in arms HPCT, ACy followed by HPCT and atezolizumab and in arm HPCT and atezolizumab
  Other Names: Perjeta
Drug: Carboplatin — Carboplatin will be given i.v. on day 1 and day 8 every 3 weeks in arms HPCT, ACy followed by HPCT and atezolizumab and in arm HPCT and atezolizumab
  Other Names: Carboplatin Hospiria
Drug: Paclitaxel — Paclitaxel will be given i.v. on day 1 and day 8 every 3 weeks in arms HPCT, ACy followed by HPCT and atezolizumab and in arm HPCT and atezolizumab
  Other Names: Paclitaxel Hospiria
Drug: Doxorubicin — Adriamycin will be delivered i.v. on day 1 every 3 weeks in arm ACy followed by HPCT for the first 3 cycles
  Other Names: Doxorubicin Pfizer
  Arms: ACy followed by HPCT and atezolizumab
Drug: Cyclophosphamide — Cyclophosphamide will be given i.v. on day 1 every 3 weeks in arm ACy followed by HPCT and atezolizumab for the first 3 cycles
  Other Names: Cyclophosphamide Sandoz
  Arms: ACy followed by HPCT and atezolizumab
Drug: Atezolizumab — Atezolizumab will be given i.v. on day 1 every 3 weeks in arm ACy followed by HPCT and atezolizumab and in arm HPCT and atezolizumab
  Other Names: Tecentriq
  Arms: ACy followed by HPCT and atezolizumab; HPCT and atezolizumab
Procedure: Surgery — Breast cancer surgery (breast and axilla) either conservative or radical not later than 4 weeks from the last dose of neoadjuvant therapy in all study arms

SUMMARY:
n the present study the neoadjuvant approach with the anti-HER2 trastuzumab and pertuzumab combined with carboplatin and paclitaxel will be used to compare the Event-Free Survival (EFS) in regimens with and without atezolizumab. Following the neoadjuvant part of the study, after surgery all patients will continue to receive trastuzumab and pertuzumab to complete one year of anti-HER2 therapy. Similarly, patients allocated to receive atezolizumab will continue atezolizumab to complete one year In addition, several IHC and molecular assays will be performed before and during the period of chemotherapy administration and at surgery with the goal of defining a marker of efficacy to be later validated in a larger adjuvant setting.

DETAILED DESCRIPTION:
Dual targeting of HER2 with trastuzumab and pertuzumab in HER2-positive breast cancer is linked to clinical evidence of reversal of initial resistance to trastuzumab (Baselga J et al, J Clin Oncol 2010) in cases progressing on trastuzumab therapy, and in dramatic improvement in progression free and overall survival when the two monoclonal antibodies are used in combination with docetaxel (THP regimen) as first line therapy of metastatic disease as shown in the CLEOPATRA study (Swain S et al, ESMO abstract 2014). The randomized NeoSphere study showed that the same THP regimen given for 4 cycles as neoadjuvant treatment increased the rate of pathologic complete response (pCR) over that with conventional docetaxel and trastuzumab or docetaxel and pertuzumab (Gianni L et al, Lancet Oncol 2012).

Encouraging clinical data emerging in the field of tumor immunotherapy have demonstrated that therapies focused on enhancing T cell responses against cancer can result in a significant survival benefit in patients with advanced malignancies (Hodi FS and Dranoff G, J Cutan Pathol 2010; Kantoff PW et al, New Engl J Med 2010; Chen DS et al, Clin Cancer Res 2012). Many human tumors have been found to overexpress PD L1, which acts to suppress anti tumor immunity. PD 1 is an inhibitory receptor expressed on T cells following T cell activation, which is sustained in states of chronic stimulation, such as in chronic infection or canc Atezolizumab is a human monoclonal antibody containing an engineered Fc-domain to optimize efficacy and safety that targets PD-L1 and blocks binding of its receptors, including PD-1 and B7.1.

In addition to being involved in the natural progression of cancer, immunity can affect the activity of various anticancer agents. Accordingly, recent evidence suggests that some chemotherapeutic drugs, such as anthracyclines and oxaliplatin, rely on the induction of anticancer immune responses. Immune responses also play a major role in the efficacy of targeted therapies with monoclonal antibodies (Stagg J et al, Breast Care 2012). Studies have shown monoclonal antibodies such as trastuzumab and rituximab rely in part on immunemediated killing through antibody-dependent cellular cytotoxicity (ADCC). While innate immune responses appear to be important for tumor antigen-targeted monoclonal antibody therapies, recent studies in mice and correlative clinical evidence suggest that trastuzumab may also stimulate adaptive antitumor immunity. These studies raise the possibility that combination strategies may be used to capitalize on the adaptive tumor-specific immunity generated by anti-HER2 monoclonal antibodies.

Based on these considerations, we plan to conduct a randomized neoadjuvant study of the combination of trastuzumab, pertuzumab, carboplatin and paclitaxel with or without atezolizumab in women with early high-risk and locally advanced HER2-positive suitable for neoadjuvant therapy. One study arm will also include anthracycline and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 years or older with early high-risk ((T1cN1; T2N1; T3N0) or locally advanced and inflammatory breast cancers (stage III A-C according to AJCC) suitable for neoadjuvant treatment
2. Histologically confirmed unilateral invasive breast cancer
3. HER2 positive disease according to ASCO/CAP guidelines 2013 [defined as IHC 3+ or ISH positive (by gene copy number or HER2 gene/CEP17 ratio of 2 or greater)]
4. Known estrogen (ER) and progesterone receptor (PgR)
5. Availability of a representative paraffin-embedded (FFPE) tumor block taken at diagnostic biopsy for central confirmation of HER2 eligibility, for assessment of ER, PgR, Ki67 and PD-L1 expression and for biomarker evaluation is mandatory. Note: the diagnostic biopsy of the breast lesion may have been taken before the required screening procedures. If diagnostic sentinel node biopsy if performed, an FFPE block must be available. An FFPE tumor block is also mandatory after the first cycle of therapy. Surgery tissue (residual tumor or tumor bed in case of pCR and axillary node material) is also mandatory.
6. Consent to the collection of blood samples mandatorily before starting neoadjuvant treatment, after the first cycle of therapy, at the end of neoadjuvant treatment (before surgery), 6 months after surgery and at the end of all treatments.
7. ECOG performance status 0 or 1
8. For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drugs. Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Examples of contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide
9. Written informed consent to participate in the trial (approved by the Institutional Review Board [IRB]/ Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures
10. Willing and able to comply with the protocol

Exclusion Criteria:

1. Evidence of bilateral breast cancer or metastatic disease (M1)
2. Patients with HER2-negative defined as 0-1+ by immunohistochemistry or 2+ by immunohistochemistry without HER2 amplification by either In Situ Hybridization (ISH) or other amplification tests done locally are considered not eligible for the study
3. Pregnant or lactating women. Documentation of a negative pregnancy test must be available for premenopausal women with intact reproductive organs and for women less than one year after the last menstrual cycle
4. Women with childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception, for example abstinence, an intra-uterine device, or double barrier method of contraception
5. Previous treatment with chemotherapy, hormonal therapy or an investigational drug for any type of malignancy
6. Previous investigational treatment for any condition other than malignancy within 4 weeks of randomization date
7. Administration of a live, attenuated vaccine within 4 weeks before Day 1 or anticipation that such a live attenuated vaccine will be required during the study
8. Previous or concomitant malignancy of any other type that could affect compliance with the protocol or interpretation of results. Patients with curatively treated basal cell carcinoma of the skin or in situ cervix cancer are generally eligible
9. Pre-existing motor or sensory neuropathy of grade > 1 for any reason
10. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
11. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
12. Patients with prior allogeneic stem cell or solid organ transplantation
13. History of autoimmune disease including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
14. History of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) or evidence of active pneumonitis on screening chest computed tomography scan
15. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
16. History of HIV infection, active hepatitis B (chronic or acute), or hepatitis C infection. Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [anti-HBc] test) are eligible.

    Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction assay (PCR) is negative for HCV RNA
17. Active tuberculosis
18. Severe infections within 4 weeks prior to Day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. Signs or symptoms of significant infection within 2 weeks prior to Day 1
19. Received oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
20. Other serious illness or medical condition including: history of documented congestive cardiac failure; New York Heart Association (NYHA) Class II or greater CHF; angina pectoris requiring anti-anginal medication or unstable angina within 6 months prior to Day 1; evidence of transmural infarction on ECG; myocardial infarction stroke or transient ischemic attack (TIA) within 6 months prior to Day 1; poorly controlled hypertension (e.g. systolic >180 mm Hg or diastolic >100 mm Hg; however, patients with hypertension which is well controlled on medication are eligible); clinically significant valvular heart disease; high-risk uncontrolled arrhythmias
21. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent or adversely affecting compliance with study drugs
22. Serious uncontrolled infections (bacterial or viral) or poorly controlled diabetes mellitus
23. Any of the following abnormal baseline hematological values:

    1. White blood count (WBC) < 2.5 x 109/L
    2. Absolute Neutrophil Count (ANC) < 1.5 x 109/L
    3. Lymphocyte count < 0.5 x 109/L
    4. Platelet count < 100 x 109/L
    5. Hemoglobin (Hb) < 10 g/dL
24. Any of the following abnormal baseline laboratory tests

    1. Serum total bilirubin > 1.5 x ULN (upper limit of normal) (except for patients with clearly documented Gilbert's syndrome)
    2. Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.25 x ULN
    3. Alkaline phosphatase > 2.5xx ULN
    4. Serum creatinine > 1.5 x ULN
    5. INR and aPTT > 1.5 × ULN within 2 weeks prior to enrollment. This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
25. Baseline left ventricular ejection fraction (LVEF) < 50% by echocardiography or multi-gated scintigraphic scan (MUGA)
26. Major surgical procedure within 28 days prior to Day 1 or anticipation of need for a major surgical procedure during the course of the study
27. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to Day 1 or at any time during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 5 years after the randomization of the last patient
  Assess EFS (disease progression while on neoadjuvant therapy or disease recurrence after surgery) in the study arms

SECONDARY OUTCOMES:
Pathological complete response (pCR) | At surgery, an expected average of 26 weeks after the randomization of the last patients
  Assess the rate of pCR defined as absence of invasive cancer in both breast and axillary nodes (ypT0Tis ypN0)
Clinical objective response | Participants will be followed for the duration of neoadjuvant therapy, an expected average of 22 weeks
  Assess the rate of clinical response rate after neoadjuvant therapy
Distant Event Free Survival (DEFS) | 5 years after the randomization of the last patients
  Assess DEFS (defined as the occurrence of distant disease progression while on neoadjuvant therapy or distant disease recurrence after surgery) in the study arms
Overall Survival (OS) | 5 years after the randomization of the last patient
  Assess OS in all arms
Number of participants with adverse events as a measure of safety and tolerability | Participants will be followed for up to 5 years from the last randomized patient
  Number of participants with adverse events and related grades in all arms

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gianni, MD, Study Chair — Ospedale San Raffaele
Locations (65):
- Austria (4):
  - Klinikum Klagenfurt am Wörthersee Abteilung für Innede Medizin und Hämatologie und internistische Onkologie, Klagenfurt
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Universitätsklinikum St. Pölten Klinische Abteilung für Innere Medizin, Sankt Pölten
  - Klinische Abteilung für Allgemeine Gynäkologie und Gynäkologische Onkologie - Universitätsklinik für Frauenheilkunde Medizinische Universität Wien / AKH ", Vienna
- Germany (17):
  - Klinik für Gynäkologie am Campus Charité Mitte (CCM), Berlin
  - Department of Gynecology and Obstetrics, Marienhospital, Bottrop
  - Klinikum Coburg, Frauenklinik, Coburg
  - St Johannes Hospital, Dortmund
  - Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe - Universitätsklinikum Carl Gustav Carus, Dresden
  - Markus Krankenhaus - Klinik für Gynäkologie und Geburtshilfe, Frankfurt
  - SRH Waldklinikum, Gera
  - Universitätsklinikum Greifswald, Frauenklinik, Greifswald
  - Klinik und Poliklinik für Gynäkologie am Universitätsklinikum (Saale), Halle
  - Gynäkologisch-Onkologische Praxis, Hanover
  - NCT Nationales Zentrum für Tumorerkrankungen Gynäkologische Onkologie, Frauenklinik, Heidelberg
  - St. Marien-Klinik GmbH Frauenklinik der St. Vincentius-Kliniken gAG - Gynäkologisches Krebszentrum Karlsruhe - Brustzentrum Karlsruhe, Karlsruhe
  - Städtisches Klinikum Magdeburg - Klinik für Allgemein - und Viszeralchirurgie, Magdeburg
  - Am Schillerhain 1-8, Marktredwitz
  - Klinikum Nürnberg Nord, Nuremberg
  - Onkologische Praxis Velbert, Velbert
  - Marien Hospital Witten, Witten
- Italy (17):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Presidio Ospedaliero Di Summa-Perrino, Brindisi
  - Dipartimento di Oncologia Medica AUSL della Romagna, Faenza
  - IST San Martino, Genova
  - Istituto Scientifico Romagnolo per lo studio e la cura dei tumori, Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Luigi Sacco, Milan
  - Ospedale San Raffaele, Milan
  - AO Universitaria Policlinico di Modena, Modena
  - Ospedale Sacro Cuore - Don Calabria, Negrar
  - Fondazione Salvatore Maugeri, Pavia
  - Azienda Ospedaliero Universitaria Pisana Ospedale S. Chiara, Pisa
  - Arcispedale Santa Maria Nuova - A.O. Reggio Emilia, Reggio Emilia
  - Ospedale Infermi AUSL della Romagna, Rimini
  - Istituto Nazionale Tumori - Regina Elena, Roma
  - Ospedale Santa Maria della Misericordia, Udine
- Spain (27):
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Virgen de Los Lirios, Alcoy
  - Hospital General Unv. Alicante, Alicante
  - "Hospital Infanta Cristina de Badajoz (CICAB - Centro de Investigación Clínica del Área de Salud de Badajoz)", Badajoz
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic Provincial, Barcelona
  - Hospital del Mar - IMAS, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Virgen de la Nieves, Granada
  - Hospital Juan Ramón Jimenez, Huelva
  - Hospital Gregorio Marañon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Unv. Fundación Jimenez Diaz, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Complejo Hospitalario de Especialidades Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Clinica Universitaria de Navarra, Pamplona
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital de Donostia, San Sebastián
  - Hospital Onkologikoa, San Sebastián
  - Hospital Clinico Unv. de Santiago, Santiago de Compostela
  - Hospital Virgen de la Salud de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No